CLINICAL TRIAL: NCT03130374
Title: Treatment of Laryngotracheal Stenosis Using Autologous Olfactory-mucosa-derived Mesenchymal Stem Cells
Brief Title: Treatment of Laryngotracheal Stenosis Using Mesenchymal Stem Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Republican Research and Practical Center for Epidemiology and Microbiology (Other)
Collaborators: Belarusian Medical Academy of Post-Graduate Education (Other); The Republican Center for Research and Practice in Otolaryngology (Unknown)
Responsible Party: Principal Investigator, Andrei Y. Hancharou, Head of the Laboratory for Immunology and Cellular Biotechnology,, The Republican Research and Practical Center for Epidemiology and Microbiology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRPCEM_MSC1
Record Dates: First submitted 2017-04-12; First posted 2017-04-26 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Tracheal Stenosis; Laryngeal Stenosis; Mesenchymal Stem Cells
Keywords: mesenchymal stem cells; Tracheal Stenosis; Laryngeal Stenosis; cell therapy
MeSH Terms: conditions — Tracheal Stenosis; Laryngostenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cell treated group (Experimental): Patients treated according to current clinical protocols plus autologous olfactory mucosa-derived mesenchymal stem cells
  Interventions: Biological: Olfactory mucosa-derived mesenchymal stem cells
- Control group (No Intervention): Patients treated according to current clinical protocols

INTERVENTIONS:
Biological: Olfactory mucosa-derived mesenchymal stem cells — Olfactory mucosa-derived mesenchymal stem cells
  Arms: Mesenchymal stem cell treated group

SUMMARY:
The trial evaluates the safety and efficacy of the olfactory mucosa-derived mesenchymal stem cells based therapy for the patients with chronic laryngeal and tracheal stenosis

DETAILED DESCRIPTION:
Trial evaluating the safety and efficacy of olfactory mucosa-derived mesenchymal stem cells based therapy for the patients with chronic laryngeal and tracheal stenosis.

Mesenchymal stem cells are obtained from tissue biopsy of olfactory mucosa using explant method. Biomass of autologous mesenchymal stem cells in 10% human albumin solution is injected submucosally around and over the tissue after removal of a granuloma tissue during surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of chronic laryngeal or tracheal stenosis;
* absence of cartilage damage.

Exclusion Criteria:

* refuse of patient to participate in the trial;
* acute infectious diseases;
* chronic mental disorders with severe manifestations;
* pregnancy/lactation;
* intercurrent severe chronic diseases;
* HIV, Hepatites B/C;
* active tuberculosis;
* alcohol use disorder/drug addiction;
* cachexia of any origin;
* malignant neoplasms.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-01-03 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Number of patients who didn't require the repeated surgical interventions | 1 year

SECONDARY OUTCOMES:
Tracheostomy decannulation | 6 month
  Removal of the tracheostomy tube after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Y Hancharou, Dr, Principal Investigator — Head of the Laboratory for Immunology and Cellular Biotechnology, The Republican Research and Practical Center for Epidemiology and Microbiology; Valery L Chekan, Dr, Study Chair — Associate Professor of the Belarusian Medical Academy of Post-Graduate Education
Locations (2):
- Belarus (2):
  - The Republican Center for Research and Practice in Otolaryngology, Minsk
  - The Republican Research and Practical Center for Epidemiology and Microbiology, Minsk

IPD SHARING:
Plan to Share IPD: No